CLINICAL TRIAL: NCT06163430
Title: A Phase 1/2 Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of TERN-701 in Participants With Chronic Myeloid Leukemia
Brief Title: A Phase 1/2 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of TERN-701 in Participants With Chronic Myeloid Leukemia (CARDINAL)
Acronym: CARDINAL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Terns, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TERN701-1012
Record Dates: First submitted 2023-11-08; First posted 2023-12-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase; Chronic Myeloid Leukemia
Keywords: allosteric inhibitor of BCR-ABL1; CML; TERN-701; chronic myeloid leukemia; T315I; T315I mutant; CARDINAL; HS-10382
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Intervention Model Description: A sequential Intervention Model was used for Part 1 Dose Escalation. In the Part 2 Randomized Dose Expansion, participants will be randomized to one of two selected doses in parallel for the duration of the study. Participants enrolled into Part 2m (mutational cohort) will receive the same selected dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1- Dose Level 1 (160 mg) of TERN-701 (Experimental): Dose Level 1 of TERN-701 dosed once daily.
  Interventions: Drug: TERN-701
- Part 1- Dose Level 2 (320 mg) of TERN-701 (Experimental): Dose Level 2 of TERN-701 dosed once daily.
  Interventions: Drug: TERN-701
- Part 1- Dose Level 3 (400 mg) of TERN-701 (Experimental): Dose Level 3 of TERN-701 dosed once daily.
  Interventions: Drug: TERN-701
- Part 1- Dose Level 4 (500 mg) of TERN-701 (Experimental): Dose Level 4 of TERN-701 dosed once daily.
  Interventions: Drug: TERN-701
- Part 2 - Dose 1 (320 mg) (Experimental): Dose 1 was selected based on the totality of safety, PK, PD and efficacy data from Part 1. TERN-701 administered once daily.
  Interventions: Drug: TERN-701
- Part 2 - Dose 2 (500 mg) (Experimental): Dose 2 was selected based on the totality of safety, PK, PD and efficacy data from Part 1. TERN-701 administered once daily.
  Interventions: Drug: TERN-701
- Part 2m - 500 mg Dose (Experimental): Dose for Part 2m was selected based on the totality of safety, PK, PD and efficacy data from Part 1 and nonclinical data. TERN-701 is administered once daily.
  Interventions: Drug: TERN-701

INTERVENTIONS:
Drug: TERN-701 — TERN-701 orally QD

SUMMARY:
The goal of the study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy of TERN-701, a highly selective allosteric inhibitor of BCR-ABL1, in participants with previously treated chronic phase - chronic myeloid leukemia (CP-CML).

The study has two parts: Part 1 of the trial (Dose Escalation) will evaluate sequential dose escalation cohorts of TERN-701 administered once daily.

Part 2 (Dose Expansion) consists of randomized, parallel dose expansion cohorts of TERN-701 that will further evaluate the efficacy and safety of 2 recommended dose levels for expansion selected from Part 1. Part 2m (mutation cohort) will further evaluate the efficacy and safety of 500mg of TERN-701 in previously treated CP-CML participants with certain resistance mutations.

In both Part 1 and Part 2, participants will receive continuous once daily dosing of TERN-701 divided into 28-day cycles. During the treatment period, participants will have scheduled visits to the trial center at Cycle 1 day 1(C1D1), C1D2 (Part 1 only), C1D8, C1D15, and C1D16 (Part 1 only), followed by Day 1 of Cycles 2 through 7, and Day 1 of every 3 cycles thereafter.

Approximately 180 participants could be enrolled in this trial, up to 80 participants in Part 1 (dose escalation), including optional backfill cohorts, approximately 80 participants in Part 2 (randomized dose expansion), and approximately 20 participants in Part 2m (mutation cohort).

All participants will receive active trial intervention.

Four dose-level cohorts have been evaluated in Part 1; two dose levels will be evaluated in Part 2 (Randomized Dose Expansion), and one dose level will be evaluated in Part 2m (mutation cohort).

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female participants ≥ 18 years of age at the time of signing the informed consent
* Have an ECOG performance status score of 0 to 2
* Have an established cytopathologically confirmed diagnosis of BCR-ABL1 positive CML in Chronic Phase
* Have received treatment with at least one prior TKI and have treatment failure, suboptimal response, or treatment intolerance
* Prior treatment with asciminib is allowed
* Adequate organ function, as assessed by local laboratory

Key Exclusion Criteria:

* Systemic antineoplastic therapy (including prior TKIs, interferon-alfa, therapeutic antibodies, chemotherapy) or other experimental therapy 7 days before the first dose of TERN-701
* Have completed previous anticancer therapy without resolution of all associated clinically significant toxicity (to ≤ Grade 2 or baseline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Part 1 - Incidence of Dose Limiting Toxicities during the first cycle of treatment | First cycle is 28 days
  Determination of the Maximum Tolerated Dose (MTD) and recommended doses for expansion cohorts of TERN-701.
Part 1 - Serious Adverse Events | up to 3 years
  Number and percentage of patients with any serious adverse event
Part 1 - Adverse Events | up to 3 years
  Number and percentage of patients with any adverse event
Part 2- Complete Hematologic Response (CHR) | up to 3 years
  CHR Defined by ELN 2020 criteria in participants who are not in CHR at baseline.
Part 2: Molecular response (MR) | up to 3 years
  MR defined by ELN 2020 criteria measured by quantitative polymerase chain reaction of BCR-ABL transcript levels.
Part 2 - Best categorical shift in BCR-ABL1 transcript levels from baseline | up to 3 years
  The best categorical molecular response shift on treatment relative to baseline

CONTACTS AND LOCATIONS:
Locations (54):
- United States (18):
  - University of Alabama Medicine (UAB Medicine), Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - UC Irvine Health, Orange, California
  - Rocky Mountain Cancer Centers, LLP, Lone Tree, Colorado
  - Florida Cancer Specialists - South Region Research Office, Fort Myers, Florida
  - Florida Cancer Affiliates - Ocala, Ocala, Florida
  - Florida Cancer Specialists - North Region Research Office, St. Petersburg, Florida
  - Florida Cancer Specialists - East Region Research Office, West Palm Beach, Florida
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Memorial Sloan Kettering Cancer Center - Main Campus, New York, New York
  - Atrium Health Levine Cancer Institute, Winston-Salem, North Carolina
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Thomas Jefferson University - Center City (Philadelphia), Philadelphia, Pennsylvania
  - Tristar BMT, Nashville, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (4):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- France (6):
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - Institut Bergonié, Bordeaux
  - Institut Paoli Calmettes, Marseille
  - CHU de Nantes (University Hospital of Nantes) - Hôtel Dieu, Nantes
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
- Germany (7):
  - Universitätsklinikum Aachen, Aachen
  - Charité Campus Virchow-Klinikum - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Mannheim, Mannheim
  - Klinikum rechts der lsar der Technischen Universität München, München
- Italy (4):
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant'Orsola, Bologna
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS San Gerardo dei Tintori - SC Centro di Ricerca Fase I, Monza
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
- South Korea (4):
  - Uijeorigbu Eulji Medical Center, Eulji University, Uijeongbu-si, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggido
  - Dong-A University hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
- Spain (8):
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitari Germans Trias i Pujol (ICO Badalona), Barcelona
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital de Día Quirónsalud Zaragoza, Zaragoza
- Imperial College Healthcare NHS Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No